CLINICAL TRIAL: NCT02316678
Title: Patient Attitudes and Preferences for Outcomes of Inflammatory Bowel Disease Therapeutics
Acronym: PPOD
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Crohn's and Colitis Foundation (Other); University of Alabama at Birmingham (Other); Duke University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, James Lewis, Professor of Medicine, University of Pennsylvania
Other Study IDs: 818347
Record Dates: First submitted 2014-12-01; First posted 2014-12-15 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Colitis, Ulcerative; Inflammatory Bowel Diseases; Crohn's Disease
Keywords: Patient Preference
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases; Crohn Disease; Patient Preference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- anti-TNF - no intervention: Patients who are new users of anti-TNF therapy
  Interventions: Other: No intervention
- Corticosteroids - no intervention: Patients initiating corticosteroids
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention

SUMMARY:
The investigators will test the hypothesis that that greater efficacy of anti-tumor necrosis factor (antiTNF) therapy results in reduced need for bowel resection surgery, fewer serious infections, and reduced short term mortality risks, and therefore has a more favorable benefit to harm profile than corticosteroids for inflammatory bowel disease.

DETAILED DESCRIPTION:
The investigators will conduct a comparative effectiveness study among Medicare Parts A, B, and D beneficiaries with inflammatory bowel disease. The investigators will compare the incidence of severe infection, bowel resection surgery, and death among new users of anti-tumor necrosis factor therapies and corticosteroids. The investigators will compute propensity scores to describe the propensity for treatment with anti-tumor necrosis factor drugs compared to corticosteroids, and will match corticosteroids and anti-tumor necrosis factor drug treated patients on the propensity score. Cox regression will be employed to assess the hazard ratio for each of the outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be required to have at least two diagnosis of inflammatory bowel disease within the 6 months prior to initiating anti-TNF therapy or corticosteroids. To assure full coverage, patients will be required to have Parts A, B, and D Medicare coverage.

Exclusion Criteria:

1. Diagnosis of rheumatoid arthritis, psoriasis, ankylosing spondylitis, or psoriatic arthritis in the 6 months period prior to initiation of the therapy.
2. Less than 6 months of follow-up time within the data source prior to initiation of the therapy.
3. Diagnosis of cancer in the 6 months prior to initiation of the study medication.
4. Initiation of anti-TNF therapies within the first 6 months following surgery.
5. Patients who are in managed care plans (Medicare Part C).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will use Medicare data from 2006-2011. Patients will be required to have at least two diagnosis of inflammatory bowel disease within the 6 months prior to initiating anti-TNF therapy or coritcosteroids as defined below. To assure full coverage, patients will be required to have Parts A, B, and D Medicare coverage.
Sampling Method: Non-Probability Sample
Enrollment: 9573 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Lewis, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Bewtra M, Reed SD, Johnson FR, Scott FI, Gilroy E, Sandler RS, Chen W, Lewis JD. Variation Among Patients With Crohn's Disease in Benefit vs Risk Preferences and Remission Time Equivalents. Clin Gastroenterol Hepatol. 2020 Feb;18(2):406-414.e7. doi: 10.1016/j.cgh.2019.05.010. Epub 2019 May 14. PMID 31100456

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a retrospective cohort study of Medicaid and Medicare beneficiaries with Inflammatory Bowel Disease (IBD) in the United States using administrative data. Medicaid data were from 2001-2005 and Medicare data were from 2006-2013.
Period: Overall Study
Arm/Group | Anti-TNF - no Intervention | Corticosteroids - no Intervention
Started | 1879 | 7694
Completed | 1879 | 7694
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti-TNF - no Intervention | Corticosteroids - no Intervention | Total
Number analyzed (Participants) | 1879 | 7694 | 9573
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1323 | 4838 | 6161
  >=65 years | 556 | 2856 | 3412
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (17.7) | 53.2 (18.8) | 52.6 (18.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1216 | 4830 | 6046
  Male | 663 | 2864 | 3527
Region of Enrollment [Number; unit: participants]
  United States | 1879 | 7694 | 9573

OUTCOME MEASURES:

1. Primary Outcome: Mortality Rate
Description: Incidence of death per 1000 person-years
  Outcome Measure Time Frame:Follow-up was from the date that the participant first met the criteria for either prolonged corticosteroid use or new anti-TNF use until either the patient died, discontinued enrollment in Medicaid or Medicare Part A, B, or D, reached age 90, was newly diagnosed with other immune-mediated diseases or AIDS, or reached the end of the available data, whichever came first, assessed up to 13 years. Follow-up of patients with UC also ended if they were diagnosed with a fistula, as this would usually change the diagnosis to CD.
Time Frame: See Outcome Measure Description above
Population: Patients treated with corticosteroids (CS) within the prior year and subsequently received either additional CS therapy meeting the definition of prolonged CS use or newly initiated anti-TNF therapy were included in the study.
Measure: Number; unit: events per 1000 person-years
Groups:
- Anti-TNF: New users of anti-TNF therapy defined as ≥ 1 dispensing for an anti-TNF drug with ≥1 filled CS prescription and no dispensing for any anti-TNF medication in the 12 months preceding the first anti-TNF dispensing.
- Steroids: Prolonged users of steroids defined as either >3000 mg of prednisone (or equivalent) or >600 mg of budesonide divided between ≥2 prescriptions within 12 months and absence of any anti-TNF therapy during the same 12 months.
Arm/Group | Anti-TNF | Steroids
Number analyzed (Participants) | 1879 | 7694
events per 1000 person-years | 21.4 | 30.1

ADVERSE EVENTS:
Arm/Group | Anti-TNF - no Intervention | Corticosteroids - no Intervention
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No